CLINICAL TRIAL: NCT06187636
Title: Pictures Of Hope: Parents Reflecting On Hope During Hospice Through Photovoice
Brief Title: Parents Reflecting On Hope During Hospice Through Photovoice
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PHOTOHOPE
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Bereavement
Keywords: Photovoice; Bereaved parent; Hospice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, researchers will use Photovoice to learn about how bereaved parents felt and thought about hope when their children were on hospice. 'Photovoice' is a research method that uses participants' photographs as a springboard for discussion.

Primary Objective

* To explore reflections, emotions, and experiences evoked in bereaved parents when reviewing photographs from their child's time on hospice, with photos selected by parents based on a prompt related to their thoughts about hope during that time.

DETAILED DESCRIPTION:
Using a prospective qualitative design, we will enroll parents of children who died on hospice 6-24 months prior. Parents who opt to participate in the study will be asked to review photographs they have from when their child was on hospice and to select 1-5 photographs that communicate what hope meant to them at that time. Their photograph selection will be guided by a brief conversation with the researcher and a written guide that encourages the participant to think about hope broadly and invites an open interpretation of what it means for a photograph to represent hope.

Parents will bring their selected photograph(s) to a one-on-one semi-structured interview. The interview will take place either in person or over a virtual meeting platform. During the interview, the participant will share the photographs with the researcher, discuss why they were chosen, and share any other reflections they have about their experience. It is anticipated that the interview will last about 60 minutes. The audio for the meeting will be recorded. Video will not be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be the parent of a child who:

  * Received any form of care from a clinician at St. Jude, as documented in the electronic medical record, AND
  * Was enrolled on hospice at the time of death, AND
  * Died at least 6 months prior to enrollment, but no more than 24 months prior to enrollment.
* Participants must also:

  * Be ≥ 18 years of age or legally emancipated, AND
  * Be English-speaking or Spanish-speaking.

Exclusion Criteria:

* Insufficient comfort or fluency with either English or Spanish language.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Those who meet the Eligibility Criteria and agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of reflections, emotions, and experiences evoked in bereaved parents when reviewing photographs from their child's time on hospice | Approximately 1- 3 weeks after enrollment (The time frame will be flexible to allow for maximal convenience to the participant, with participants empowered to select an interview date outside of the timeframe at their discretion.)
  The unit of analysis will be the semi-structured interview, including the transcript and any field notes taken by the researcher during or immediately after each interview. Interviews will be recorded, transcribed, de-identified, and analyzed using qualitative inductive content analysis. Content analysis will include memo-writing, codebook development, coding, reconciliation, and synthesis to identify meaningful patterns and themes. MAXQDA, a sophisticated qualitative analysis software system, will be used to conduct and synthesize analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Superdock, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols